CLINICAL TRIAL: NCT01593176
Title: Radiostereometric Analysis of Fracture Healing in Distal Femur Fractures
Acronym: RSA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Mark Steven Vrahas, Chief, Orthopaedic Trauma Service, Massachusetts General Hospital
Other Study IDs: 2011P001012
Record Dates: First submitted 2012-05-02; First posted 2012-05-08 (Estimated); Last update posted 2015-05-06 (Estimated); Status verified 2015-05

CONDITIONS: Distal Femur Fractures
Keywords: Femur; Fracture; Radiostereometric Analysis
MeSH Terms: conditions — Femoral Fractures, Distal; Fractures, Bone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Distal Femur Fracture, LISS Plate: Patients presenting with a distal femur fracture requiring surgical fixation with a Less Invasive Stabilization System (LISS) plate will have placement of RSA beads for analysis.
  Interventions: Procedure: Placement of RSA beads

INTERVENTIONS:
Procedure: Placement of RSA beads — At the time of surgery sets of up to 9 RSA beads will be implanted on sides of the main fractures lines with the use of the inserter instrument and the image intensifier. In AO/OTA type 33A fractures two sets will be implanted - one in the femoral shaft and one in the distal femoral epiphysis. In AO/OTA type 33C fractures with an extra fracture line through the epiphysis, three sets will be implanted - one in the femoral shaft, one in the main lateral condyle segment and one in the main medial condyle segment. No beads will be planted in comminuted bone fragments. The fracture will then be plated with a LISS plate as it normally would.
  Other Names: RSA Biomedical Tantulum Markers; Synthes Less Invasive Stabilization System Fixation Plate

SUMMARY:
The investigators are doing this research study to look at how distal femoral fractures (knee bone break) heal. In this study, the investigators will use Radiostereometric Analysis (RSA) to look at how the pieces of femur bone move as the bone heals. RSA is a special x-ray that uses radiographs to measure very small movements in the bone over time. The question that will be answered by this study is whether RSA can be used as a tool to monitor fracture healing.

DETAILED DESCRIPTION:
Determining when a fracture has united can be very difficult. Plain radiographs are easy to obtain but are notoriously inaccurate for determining union. CT scans are more helpful, but are more costly and inconvenient. Artifacts from the metal implants often mask the visibility of the bone structure. In addition, the accuracy of CT scans for determining non-unions is not known. CT scanning will identify a nonunion when a clear persistent fracture line separates the fragments. Unfortunately, the scans often reveal some areas where bone has bridged the fracture, and other areas where the fracture line remains. Ultimately, no one knows the amount of bridging necessary to stop motion between the fragments. Often the best indication of fracture healing is the resolution of pain. However, patients' pain tolerance varies greatly. It is clear that our specialty needs better techniques to determine fracture union. This is particularly important since the market is introducing many new drugs that purport increased rate of fracture healing. If there are no standards to evaluate fracture healing, there is no way to determine drug efficacy.

Radiostereometric analysis (RSA) is a highly accurate, precise, safe and objective technique that uses radiographs to measure very small displacements and relative motion over time. It has been used successfully for some time to evaluate small changes in the position of prosthetic joints. There is some indication that this technique can also be used to evaluate healing by determining when motion between the fragments stops. A limited number of phantom model RSA in-vitro studies have proven useful for measuring the rigidity of different types of osteosyntheses methods. However, RSA has so far only been applied in a few in-vivo studies to evaluate fracture healing.

Osteosynthesis of distal femur fractures is challenging. Fractures are reduced through a large skin incision and often patients face non-union or union in a varus or valgus deformity after a long convalescence. That said, increased fracture fixation is now achievable through the newly invented locked angle screw plate system. The Synthes product, Less Invasive Stabilization System (LISS) plate is one example of this new system. The exact time of fracture healing, however, remains uncertain. No RSA in-vivo studies have been published among patients with distal femur fractures - but one RSA in-vitro study on 18 phantom distal femurs demonstrates RSA to be a relatively simple way to collect and analyze the relative motion between fragments fixed with the LISS.8 Given this, it should be possible to evaluate fragment motion in distal femur fractures stabilized using the LISS plate in order to evaluate healing.

At the time of surgery, sets of up to 9 RSA beads will be implanted on sides of the main fractures lines with the use of the inserter instrument and the image intensifier. In AO/OTA type 33A fractures, two sets will be implanted - one in the femoral shaft and one in the distal femoral epiphysis. In AO/OTA type 33C fractures with an extra fracture line through the epiphysis, three sets will be implanted - one in the femoral shaft, one in the main lateral condyle segment and one in the main medial condyle segment. No beads will be planted in comminuted bone fragments. Patients will be evaluated during outpatient follow-up visits standard for this fracture (2 weeks, 6 weeks, 3 months, 6 months and 1 year after surgery.)

The purpose of this study is to use RSA to evaluate fracture healing in distal femoral fractures osteosynthezed using the LISS.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged 18 and older
* Isolated distal femur fracture requiring surgical stabilization with a LISS plate
* Subjects who are able to return to MGH for follow-up during the year following their injury.

Exclusion Criteria:

* Subjects with expected limited life span less than a year.
* Subjects who were non ambulatory prior to their injury
* Female subjects who are pregnant
* Subjects who are treated with an orthopaedic implant other than the LISS
* Subjects with bone structure illnesses.
* Pathologic fractures secondary to neoplasm
* Subject with a severe open distal femur fracture with vascular damage
* Subjects who are unable to attend post-operative outpatient appointments at the MGH

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All potential subjects will be in the inpatient setting of Massachusetts General Hospital or Brigham & Women's Hospital at the time of recruitment awaiting surgery on their distal femur fracture
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2012-05; Primary Completion 2015-05 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Change in inter-fragmentary motion throughout the course of healing for distal femoral fractures. | Change in inter-fragmentary motion from baseline at 2 weeks, 6 weeks, 3 months, 6 months and 1 year postoperatively
  Use radiostereometric analysis to measure inter-fragmentary motion

CONTACTS AND LOCATIONS:
Overall Officials: Mark S Vrahas, MD, Principal Investigator — Massachusetts General Hospital; Charles Bragdon, Ph.D, Principal Investigator — Massachusetts General Hospital; Michael J Weaver, MD, Principal Investigator — Brigham and Women's Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham & Women's Hospital, Boston, Massachusetts